CLINICAL TRIAL: NCT02279017
Title: Mobile Health Messages to Sustain Recent Weight Loss - Phase 2
Brief Title: mHealth Messages to Sustain Recent Weight Loss - Phase 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00057562
Record Dates: First submitted 2014-10-28; First posted 2014-10-30 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2016-03

CONDITIONS: Weight Loss
Keywords: Mobile Technology; Diet and Fitness
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Weight Loss (Other): We will send the study participate a daily text message for 2 months to their phone at 8 A.M. and a weekly text message for 6 months asking them to report their weight through a 2-question online survey. After that, a monthly text message for 18 months asking them to report their weight.
  Interventions: Behavioral: mHealth Texting for Weight Loss

INTERVENTIONS:
Behavioral: mHealth Texting for Weight Loss

SUMMARY:
To assess the feasibility to translate an automated weight loss message intervention to a weight loss clinic population.

Aim 1: To assess feasibility of translating the intervention in a clinic for patients who recently completed a structured weight loss program.

Aim 2: To assess the ability to capture a trajectory of self-reported weight over 6 months through an automated intervention.

DETAILED DESCRIPTION:
The investigators will recruit 100 participants who are clients at the Duke Diet and Fitness Center. At baseline the investigators will collect demographic information such as, their age, weight, education. When participants complete their respective program at the DFC they will receive a daily weight loss sustaining text message at 8:00 A.M. for 60 days. Participants will also receive weekly messages for 6 months asking them to self-report their weight. Thereafter, they will receive an automated message monthly for 18 months asking them to self-report their weight.

ELIGIBILITY:
Inclusion Criteria:

* A client of Duke diet and Fitness Center (DFC)
* Are able to speak and read English
* Should complete a diet and fitness program at the DFC.
* Client should own a mobile smart phone to personally receive text messages.
* Client should have access to a web-based survey to self-report their weight.

Exclusion Criteria:

* No exclusions

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Subject's weight loss | 2 years
  The study is being done to asses the ability to translate an automated weight loss message intervention to a weight loss clinic population.
Percentage of subjects who self-report weight to the clinic | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Shaw, RN, Phd, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Diet and Fitness Center, Durham, North Carolina, United States